CLINICAL TRIAL: NCT02507804
Title: A Single Centre Randomised Controlled Study to Evaluate a Diary for Patient Reported Outcome Measures (PROMs)
Brief Title: A Study to Evaluate a Diary for Patient Reported Outcome Measures (PROMs)
Acronym: PROMs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Christie NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CFTSp099
Record Dates: First submitted 2015-07-10; First posted 2015-07-24 (Estimated); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A diary arm (Experimental): Patients in Arm A are required to complete a patient diary. This will be reviewed by an Investigator at every visit in order to gain Adverse Event and Concomitant Medication information.
  Interventions: Other: Patient diary PROMs
- Arm B standard of care (Active Comparator): Patients will be asked to recall Adverse Events and Concomitant Medication information as standard of care practice would dictate.
  Interventions: Other: Counselling

INTERVENTIONS:
Other: Patient diary PROMs
  Arms: Arm A diary arm
Other: Counselling
  Arms: Arm B standard of care

SUMMARY:
The aim of the study is to design and evaluate a PROMs diary for cancer patients to self report side effects and experiences of their treatment, and thereby create a detailed account of treatment related adverse events and their impact on daily activities to share with the care team.

DETAILED DESCRIPTION:
This is a randomised, controlled, single-centred study to compare the quality of Adverse Events (AE) and Concomitant Medication (CM) reporting, patient satisfaction, care experience and quality of life in cancer patients undergoing chemotherapy and managed with/without a diary for Patient Reported Outcome Measures.

164 subjects will be enrolled and randomised in a 1:1 ratio and stratified by line of therapy (first line vs second line or higher line), treatment intent (curative vs palliative) and ECOG performance status (0-1 vs 2-3).

All subjects will receive standard chemotherapy delivered as per institutional practice. They will also receive counselling on monitoring and reporting side effects, medication and experiences as per standard practice.

All subjects will complete a study questionnaire and EQ-5D forms in the Outpatient Department prior to the consultation and delivery of chemotherapy.

Subjects randomised to Arm A will use the PROMs diary to record side effects, medication and experiences associated with cycles 1-6 of chemotherapy. The diary will be reviewed by the study team to collect AE and CM information. AE/CM will be recorded in source documents as per usual practice.

Subjects randomised to the control Arm B will discuss side effects, medication and experiences associated with cycles 1-6 of chemotherapy at clinical consultations as per standard practice. This may include the use of notes, diaries or other methods at their own discretion. Arm B subjects may not use a PROMs diary. The study team will collect and record AE/CM information in the source documentation as per usual practice.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18 or over; no upper age limit.
* Cancer requiring commencement of chemotherapy (any line) with a regime containing at least 6 cycles (of any cycle duration).
* Chemotherapy may include any systematic anti-cancer therapy (i.e. cytotoxic agents, immunotherapy or targeted therapy) provided this is delivered as induction therapy.
* Expectation to complete cycles 1 through 6 of planned therapy.
* The capacity to understand the Patient Information Sheet and provide written informed consent.
* Non English speaking patients may enter the study if an English speaking friend or relative is willing to assist the patient.
* Willingness and ability to comply with study procedures.
* A patient enrolled on a concurrent IMP clinical trial is permitted at the Investigators discretion.

Exclusion Criteria:

* Patients who have already commenced therapy for their current disease episode i.e. received at least their first cycle of chemotherapy.
* Patients receiving chemotherapy/ radio-immunotherapy as the sole modality of treatment.
* Patients who have completed induction therapy and due to commence maintenance therapy.
* Uncontrolled medical condition that in the opinion of the Investigator may jeopardise completion of 6 cycles of treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2019-06-03 (Actual); Study Completion 2019-06-03 (Actual)

PRIMARY OUTCOMES:
adverse event and concomitant medication reporting in patient case notes as standard of care | Over 6 cycles of chemotherapy/treatment (approximately 18 weeks)

SECONDARY OUTCOMES:
Measure quality of life questionnaire (EQ5D ) | Over 6 cycles of chemotherapy/treatment (approximately 18 weeks)
Measure patient satisfaction questionnaire | Over 6 cycles of chemotherapy/treatment (approximately 18 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Kim Linton, MBChP MRCP PhD, Principal Investigator — Christie NHS Foundation Trust
Locations (1):
- Christie NHS Foundation Trust, Manchester, United Kingdom